CLINICAL TRIAL: NCT06057506
Title: Comparative, Monocentric Study for the Evaluation of the Efficacy of Two Medical Devices on the Treatment of Head Lice Infestation
Brief Title: Comparative Study for the Evaluation of Two Medical Devices on the Treatment of Head Lice Infestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Perrigo CSCI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22E1852
Record Dates: First submitted 2023-08-30; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Head Lice Infestation
Keywords: Head Lice Infestation; Pediculosis capitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Device (Experimental): Medical device for the treatment of head lice infestation: Paranix® Shampoo, already in the market in Europe
  Single topical application administered to hair and scalp for 10 minutes. Applied by principal investigator on site.
  Interventions: Device: Paranix® Shampoo
- Comparator Device (Active Comparator): Medical device for the treatment of head lice infestation: Paranix® Lotion, already in the market in Europe
  Single topical application administered to hair and scalp for 10 minutes. Applied by principal investigator on site.
  Interventions: Device: Paranix® Lotion

INTERVENTIONS:
Device: Paranix® Shampoo — well established medical device for the treatment of head lice infestation (osmolone based)
  Arms: Investigational Device
Device: Paranix® Lotion — well established medical device for the treatment of head lice infestation (dimethicone based)
  Arms: Comparator Device

SUMMARY:
Pediculosis capitis or head lice infestation is a human medical condition caused by the infestation of the hair by the parasitic insect Pediculus humanus capitis (human head lice). The most common symptom of infestation is pruritus (itching) on the head which normally intensifies 3 to 4 weeks after the initial infestation.

The test items have been developed with the ambition to offer a complete head lice treatment, whilst also offering ultimative convenience in use - making treatment of head lice infestation easy, and effective in few minutes.

The main objective of this clinical study is to confirm the efficacy on head lice treatment of two Medical Devices, already in market.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject;
* Sex: male or female;
* Age: 2 years and above;
* Subject with a slight to moderate lice infestation (according to EU norms);
* Subjects with various hair type (from 1 to 3C - hair scale) and hair length (from short to mid length hair, not exceeding shoulder);
* Documented oral informed consent for all subjects, including minors, given freely and expressly before the start of the study;
* Written informed consent for subjects ≥18 years or legal guardian for subjects < 18 years given freely and expressly before start of the study;
* Written assent for subjects ≥12 to <18 years;
* Subject/Subject's legal guardian is psychologically able to understand the study related information and to give written informed consent;
* Females of childbearing potential must have a negative pregnancy test before the beginning of the study.

Exclusion Criteria:

* Pregnant (confirmed by pregnancy test for women of childbearing potential) or nursing woman or planning a pregnancy during the study;
* Subject who had been deprived of their freedom by administrative or legal decision or adult subject who is under guardianship;
* Subject in a social or sanitary establishment;
* Subject in an exclusion period from a previous study or who is currently participating in another study on hair/scalp or who participated to another clinical study on hair/scalp within 3 months before first visit;
* Subject suspected to be non-compliant according to the investigator's judgment;
* Subject with curly or frizzy hair (from 4A to 4C in the hair type scale);
* Subject with hair length below the shoulder;
* Subjects with more than 24 lice on the head.

In terms of associated pathology

* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results;
* Subject with a cutaneous disease on the studied zone (scalp and hair);
* Subject with severe scratches or open wounds/skin damages on the scalp (lice bites allowed however);
* Subject with a known or suspected allergy to any of the components/materials of the investigational devices, anti-lice comb or post-treatment shampoo;
* Subject who has diabetes (type 1 or 2);
* Subject with known or suspected immune deficiency or autoimmune disease.

Relating to previous or ongoing treatment

* Subject undergoing a topical treatment on the test area or a systemic treatment with:

  * anti-inflammatory medication and/or anti-histamines during the previous 2 weeks and during the study;
  * corticosteroids during the 2 previous weeks and during the study;
  * retinoids and/or immunosuppressors during the 3 previous months and during the study;
  * any medication stabilized for less than one month.
* Subject who received an anti-lice treatment in the previous 2 months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy based on the cure rate after complete treatment | Day 7, Day 14 if applicable
  The cure rate is defined as the rate of subjects having no live lice on hair 7 days after the last application of the product (Day 7 or Day 14 if second application is needed).

SECONDARY OUTCOMES:
Cure rate of each individual investigational device | Day 7, Day 14
  Evaluate the cure rate of each individual investigational device
Cure rate after one dose of investigational device application | Day 7
  Comparison of the percentage of subjects cured after one dose of the investigational device compared to the percentage of subjects cured with one dose of the comparator device.
Dead and live lice/nymphs after combing | Day 0, Day 7 if applicable
  Number of dead and live lice/nymphs collected on the anti-lice comb after treatment.
Live lice and nymphs after application | Day 1, Day 7, Day 8 if applicable, Day 14 if applicable
  Evaluation of the presence of live lice and nymphs, for both groups, without combing on hair and close to scalp
Number of participants with treatment-related adverse events, serious adverse events as assessed by investigator | Day 0, Day 1, Day 7, Day 8 if applicable, and Day 14 if applicable
  Evaluation of the safety and tolerability of the investigational device versus comparator
Subject reported perceived acceptability, efficacy and subjective evaluation assessed via questionnaire | Day 1, Day 7 or Day 14 if applicable
  Evaluation of the perceived acceptability, subjective efficacy and risk of re-infestation;
  Subject perception questionnaire with the following scale items:
  totally agree, agree, rather disagree, disagree

CONTACTS AND LOCATIONS:
Overall Officials: Aslham Doarika, PhD, Principal Investigator — Insight Collective
Locations (1):
- Insight Research, Quatre Bornes, Mauritius

IPD SHARING:
Plan to Share IPD: No